CLINICAL TRIAL: NCT00692003
Title: A Double-blind, Randomised, Placebo-controlled Multi-centre Study to Assess the Efficacy and Safety of Adjunctive Zonisamide in Primary Generalised Tonic Clonic Seizures
Brief Title: Adjunctive Zonisamide in Primary Generalised Tonic Clonic Seizures
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2090-E044-315; Eudra ID #2007-003557-91.
Record Dates: First submitted 2008-06-03; First posted 2008-06-06 (Estimated); Results first posted 2012-10-12 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-02

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Zonisamide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Zonisamide (Active Comparator)
  Interventions: Drug: Zonisamide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zonisamide — 25-400 mg capsules orally once daily in the evening.
  Maximum study duration of 28 weeks comprising:
  Baseline Period (Week-8/-4 to Week 0) no treatment
  Titration Period (Week 0 to Week 4) <12 years old: 1 mg/kg; >= 12 years old: 50 mg daily titrated weekly until a dose of 5 mg/kg or 300 mg was reached by Week 4
  Maintenance Period (Week 4 to Week 16) dose from Week 4 to be maintained (4 mg/kg or 200 mg in the event of dose limiting adverse events)
  Down Titration Period (4 weeks)
  Other Names: Zonegran
  Arms: Zonisamide
Drug: Placebo — 25-400 mg Zonisamide Placebo capsules orally once daily in the evening.
  Maximum study duration of 28 weeks comprising:
  Baseline Period (Week-8/-4 to Week 0) no treatment
  Titration Period (Week 0 to Week 4) <12 years old: 1 mg/kg Zonisamide Placebo; >= 12 years old: 50 mg Zonisamide Placebo capsules daily titrated weekly until a dose of 5 mg/kg or 300 mg was reached by Week 4
  Maintenance Period (Week 4 to Week 16) dose from Week 4 to be maintained (4 mg/kg or 200 mg in the event of dose limiting adverse events)
  Down Titration Period (4 weeks)
  Arms: Placebo

SUMMARY:
Zonisamide is already marketed for the treatment of partial seizures in epilepsy. This study is intended to provide evidence that zonisamide is safe and effective in the treatment of primary generalised tonic-clonic seizures. The total trial duration will be 5.5-6.5 months. After that subjects who have completed the study will be eligible to enrol in an open-label extension study until zonisamide is marketed for this indication or further development in this indication stops. This extension study will be described in a separate protocol (E2090-E044-316).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female and aged 6-65 years.
2. Subject has ≥ 3 PGTCS over the two months before screening and during the eight weeks Baseline Period with at least one seizure in each one month period. PGTCS must occur in the context of Idiopathic Generalized Epilepsy (IGE) and may be accompanied by other primary generalized seizures, provided these are also consistent with a diagnosis of IGE.
3. Subject (or parent/caregiver, for subjects below the age of consent) is willing to sign an informed consent form. For subjects below the age of consent in their country, where appropriate they must be willing to give informed (written or verbal) assent. Subjects from the age specified in local regulations will be required to sign an appropriate informed consent form.
4. Subject is taking a stable regimen of one or two other Antiepileptic Drugs (AEDs) for at least two weeks prior to Visit 1 (start of the Baseline Period).
5. Subject has a clinical diagnosis of any type of idiopathic generalized epilepsy which has PGTCS (and which may be accompanied by other generalized seizure types), according to the International League Against Epilepsy (ILAE) Classification of Epileptic Seizures (1981) and the ILAE Classification of Epilepsies and Epileptic Syndromes (1989). Diagnosis should have been established by clinical history, electroencephalogram (EEG) and computed tomography/magnetic resonance imaging (CT/MRI) of the brain consistent with idiopathic generalized epilepsy. CT/MRI scan should have been performed within five years of the screening visit or, if not available from this period, should be performed in the Baseline Period.
6. EEG should have been performed within one year of the screening visit or, if not available from this period, should be performed in the Baseline Period.
7. Female subjects are pre-menarchal, or if of childbearing potential, are not pregnant or lactating or are post-menopausal.
8. Female subjects of childbearing potential must abide by the one of the following medically acceptable contraceptive measures: oral contraception pill, contraceptive injections, implants or patches, intrauterine device in place for at least three months or vasectomised partner or abstinence throughout the study.
9. Subject has a body weight ≥ 20 kg.

Exclusion Criteria:

1. Subject has progressive or focal neurological disease (as determined by pre-existing brain imaging such as CT or MRI performed maximally five years before the screening visit), or clinically significant organic disease.
2. Subject has a history of, or results of clinical investigations (including EEG data) that are suggestive of, partial seizures as defined by the ILAE, including generalized tonic clonic seizures which are suspected to be secondarily generalized.
3. Subjects with cryptogenic or symptomatic generalized epilepsy.
4. Subjects with psychogenic seizures.
5. Subject has a history of status epilepticus within a year of screening while complying with AEDs.
6. Subject has seizures that only occur in clustered patterns.
7. Subject has a history of renal calculi or renal insufficiency (above the upper normal limits of creatinine).
8. Subject has a known diagnosis of human immunodeficiency virus (HIV) or hepatitis B or C.
9. Subject had a predisposing condition that might interfere with absorption, distribution, or excretion of zonisamide.
10. Subject has a history of sensitivity to sulfonamide drugs or zonisamide and its excipients.
11. Subject has a recent history of excessive alcohol use or drug abuse.
12. Subject has a history of suicide attempt in the five years before the screening visit..
13. Subject has abnormal screening laboratory values that were clinically significant.
14. Subject has a history of demonstrated non-compliance with treatment or the subject or parent/caregiver can be reasonably expected not to be compliant with study procedures or to complete the study.
15. Subject has participated in a study of an investigational drug or device within 30 days prior to screening.
16. Subject has received previous treatment with zonisamide.
17. Subject is treated with ketogenic diet or vagus nerve stimulator.
18. Subject has a history of necessary treatment with rescue benzodiazepines which is foreseen to continue during the study. Rescue benzodiazepines will not be allowed in this study (stable dosing with a benzodiazepine as (one of the) baseline anti-epileptic drug(s) is allowed).
19. Current psychosis or moderate to severe depression, or use of anti-psychotic drugs, MAOIs, tricyclic antidepressants, benzodiazepine or barbiturate treatment for disorders other than epilepsy, and stimulants (amphetamine derivatives) within 28 days before the screening visit.
20. Concomitant use of acetazolamide, carbonic anhydrase inhibitors such as topiramate and drugs with anticholinergic activity.
21. Concomitant use of felbamate or use of felbamate within two months prior to Visit 1.
22. Subject is not able to swallow capsules.
23. Subject is not in general good health as determined by medical history, physical exam and screening laboratory results.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-08-01 (Actual); Primary Completion 2008-11 (Actual); Study Completion 2009-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rob Van Maanen, Study Director — Eisai Limited
Locations (72):
- Australia (5):
  - Strategic Health Evaluators Pty Ltd, Chatswood, New South Wales
  - The Prince of Wales Hospital, Randwick, New South Wales
  - Austin Health, Heidelburg, Victoria
  - The Royal Melbourne Hospital, Melbourne, Victoria
  - St. Vincents Hospital, Melbourne
- Croatia (3):
  - CH Split, Split, HR
  - CH Sestre Milosrdnice University Hospital, Zagreb, HR
  - UHC Zagreb, Zagreb, HR
- Czechia (7):
  - Neurologicke oddeleni, Hradec Králové
  - Private Neurologi Office, Kroměříž
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice s poliklinikou Ostrava, Ostrava
  - Fakultni nemocnice Plzen, Pilsen
  - Nemocnice Na Homolce, Prague
  - Centrum neurologicke pece, Rychnov nad Kněžnou
- Estonia (3):
  - West-Tallinn Central Hospital, Tallinn
  - Neurodiagnostica AP OY, Tallinn
  - Tartu University Hospital, Tartu
- Finland (2):
  - Kuopio Epilepsy Center, Kuopio, SF
  - Oulu University Central Hospital, Oulu
- Germany (5):
  - Institut fur Diagnostik der Epilepsien, Berlin
  - Neurochirurgische Klinik der Universitat Freiburg, Freiburg im Breisgau
  - Interdisziplinares Epilepsiezentrum am Klinikum der Philipps-Universitat Marburg, Marburg
  - Neurologische Gemeinschaftspraxis, München
  - Universitatsklinikum Ulm, Ulm
- Hungary (9):
  - National Institute of Psychiatry and Neurology, Budapest
  - Heim Pal Hospital, Budapest
  - Szent Istvan Hospital, Budapest
  - Orszagos Idegsebeszeti Tudomanyos Intezet, Budapest
  - Bethesda Hospital for Children, Budapest
  - Bekes County Pandy Kalman Hospital, Gyula
  - Bacs-Kiskun County ONK Hospital, Kecskemét
  - Vas County Markusovszky Hospital, Szombathely
  - Veszpem County Csolnoky F. Hospital, Veszpem
- Lithuania (3):
  - Kaunas Medical University Hospital, Kaunas
  - Neuromeda, Kaunas
  - Vilnius University Hospital Santariskiu klinikos, Vilnius
- Poland (6):
  - Niepubliczny ZOZ KENDRON, Bialystok
  - Wojewodzki Szpital Specjalistyczny im. M. Kopernika, Gdansk
  - Specjalistyczny Szpital Wieloprofilowy, Katowice
  - Centrum Neurologii Klinicznej, Krakow
  - Szpital im. M. Kopernika, Lodz
  - Uniwersytet Medyczny, Poznan
- Romania (7):
  - Spitalul Clinic de Psihiatrie, Bucharest
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Centrul Medical Sana, Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta Sf Spiridon Iasi, Iași
  - Spitalul Clinic de Urgenta Sfanta Treime, Iași
  - Spitalul Clinic Judetean de Urgenta Tg Mures, Tg Mures
- Russia (11):
  - GOU VPO Krasnoyarskaya State Medical Academy of Roszdrav, Krasnoyarsk
  - FGU Moscow Research Institute of Psychiatry of Roszdrav, Moscow
  - GOU VPO Russian State Medical University of Roszdrav, Moscow
  - GOU VPO Smolensk State Medical Academy of Roszdrav, Moscow
  - GOU VPO Moscow State University of Medicine and Dentistry of Roszdrav, Moscow
  - GOU VPO Novosibirsk State Medical University of Roszdrav, Novosibirsk
  - GU St. Petersburg Research Institute of Psychoneurology, Saint Petersburg
  - St. Petersburg State Medical Pediatric Academy, Saint Petersburg
  - GOU VPO St. Petersburg State Medical University, Saint Petersburg
  - GOU VPO Smolensk State Medical Academy of Roszdrav, Smolensk
  - Yaroslavskaya State Medical Academy, Yaroslavl
- Serbia (4):
  - Clinical Center of Serbia, Belgrade
  - University Medical Center Zvezdara, Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - Clinical Center of Nis, Niš
- Ukraine (7):
  - Tsentr Psihosomatychnoyi Patologiyi Dnipropetrovskoyi oblasnoyi klinichnoyi likarni imeni Mechnikova, Dniepropetrovsk
  - Derzhavna Ustanova Institut Nevrologiy, Kharkiv
  - Kyiv City Psychiatric Hospital #2, Poliklinichne Viddilenya, Kyiv
  - Miska Klinichna psihonevrologichna Tsentr Epilepsiyi, Kyiv
  - Lvivskyiy oblasnyi Protyepileptuchnyy tsentr, Lviv
  - Odesskyy Derzhavnyy Medychnyy Universitet, Odesa
  - Vinnitskyy Natsionalnyy Medychnyy Universitet, Vinnitsa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 6 centers (3 in Romania and 1 in Australia, Hungary, and Lithuania) during the period of 01 August 2008 to 28 January 2009.
Pre-assignment Details: Twenty-one subjects were screened and 14 participants did not continue the study after screening. Seven participants entered the study but 1 participant did not receive any treatment. Consequently, 6 participants were enrolled and treated during the study. None of the 6 subjects completed treatment & all discontinued due to the Sponsor's decision.
Period: Overall Study
Arm/Group | Zonisamide | Placebo
Started | 5 | 1
Completed | 0 | 0
Not Completed | 5 | 1
Not completed — Sponsor Decision | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Zonisamide: 25-400 mg capsules orally once daily in the evening.
  Maximum study duration of 28 weeks comprising:
  Baseline Period (Week-8/-4 to Week 0) no treatment
  Titration Period (Week 0 to Week 4) <12 years old: 1 mg/kg;
  >= 12 years old: 50 mg daily titrated weekly until a dose of 5 mg/kg or 300 mg was reached by Week 4
  Maintenance Period (Week 4 to Week 16) dose from Week 4 to be maintained(4 mg/kg or 200 mg in the event of dose limiting adverse events)
  Down Titration Period (4 weeks)
- Total: Total of all reporting groups
Arm/Group | Zonisamide | Placebo | Total
Number analyzed (Participants) | 5 | 1 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (18.66) | 27.0 (NA) — N=1 | 36.5 (17.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 2 | 1 | 3

OUTCOME MEASURES:

1. Secondary Outcome: Absolute Change From Baseline in 28-day PGTC Seizure Frequency
Description: Absolute Change from Baseline in 28-day PGTC Seizure Frequency was assessed both for the Maintenance Period alone (Week 4 to Week 16) and for the entire double-blind treatment period (Week 0 to Week 16). Due to early termination of the study by the Sponsor, no formal analyses were conducted.
Time Frame: Baseline and up to 16 weeks
Population: Due to early termination of the study by the Sponsor, no formal analyses were conducted.
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Number of Participants Considered Responders as Assessed During the Maintenance Period
Description: The number of participants who were considered responders during the 12 week Maintenance Period (Week 4 to Week 16). A responder was defined as a participant with a decrease from baseline in Primary Generalised Tonic-Clonic Seizures (PGTCS) frequency of >= 50% (i.e. 28-day PGTC seizure frequency in the period from Week 4 to the Week 16 visit compared to Week -8/-4 to randomization at Week 0). Each participant's response to treatment was assessed on the basis of their seizure diaries. The diary was dispensed at the Screening Visit and maintained by the participant (parent/caregiver) through out the titration and maintenance treatment periods until the Early termination Visit at Week 16. Due to early termination of the study by the Sponsor, no formal analyses were conducted.
Time Frame: Baseline (Week -8/-4 to Week 0) and Maintenance Phase (Week 4 to Week 16)
Population: Due to early termination of the study by the Sponsor, no formal analyses were conducted.
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for approximately 3 months
Arm/Group | Placebo | Zonisamide
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/5
Other Adverse Events (participants affected / at risk) | 0/1 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=1) | Zonisamide (N=5)
Fatigue (General disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Postictal headache (Nervous system disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
This study was terminated early at the Sponsor's discretion. When this study was discontinued, only 6 subjects had been treated. Data from the 5 subjects treated with zonisamide were insufficient to draw firm conclusions regarding efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No